CLINICAL TRIAL: NCT06190223
Title: Anatomic Single Bundle Anterior Cruciate Ligament Reconstruction With a Press-fit Tibial Fixation Technique Using Periosteal - Patellar Tendon - Bone Autograft
Brief Title: Anterior Cruciate Ligament Reconstruction With a Periosteal - Patellar Tendon - Bone Autograft - The Kocabey Press-Fit Technique
Status: Recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Collaborators: Konya City Hospital (Other); Baltalimani Bone Diseases Research and Training Hospital (Other Government); Ataturk University (Other); Karadeniz Technical University (Other); Ankara Etlik City Hospital (Other Government); Fatih Sultan Mehmet Training and Research Hospital (Other); Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Enejd Veizi, MD, Assistant Professor, Ankara City Hospital Bilkent
Other Study IDs: E2-23-5650
Record Dates: First submitted 2023-11-28; First posted 2024-01-05 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: Anterior cruciate ligament rupture; Press-fit fixation; Patellar tendon graft
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Plastic Surgery Procedures; Polypyrimidine Tract-Binding Protein; Transplantation, Autologous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PPTB Group: Patients will undergo anterior cruciate ligament reconstruction with the novel PPTB graft and a tibial press-fit technique.
  Interventions: Procedure: Anterior cruciate ligament (ACL) reconstruction with a periost-patellar-tendon-bone (PPTB) autograft and a tibial press-fit technique

INTERVENTIONS:
Procedure: Anterior cruciate ligament (ACL) reconstruction with a periost-patellar-tendon-bone (PPTB) autograft and a tibial press-fit technique — A longitudinal incision will be performed starting from the central part of the patella. A ruler will be used to mark a tendon thickness of 10mm from the middle of the patellar tendon. Superiorly, the patellar periosteum will be marked with a length of 30-40mm and a width of 10mm. Inferiorly, the tibial tubercle will be marked in a trapezoidal shape with a length of approximately 35mm, a superior narrow base of 10mm and an inferior wider base of 12mm. After extraction, the superior part of the graft will be prepared with reinforced sutures in a whipstitch pattern, while the bone block will be shaped according to the planned tunnel width. After adequate preparation, the femoral end of the graft will be shuttled in with an adjusted fixation device, while the tibial end will be hammered in with a small mallet, in a press-fit fashion, stopping short of the joint surface, but tensioned appropriately. The femoral adjustable device will then be tensioned to ensure proper graft sitting.

SUMMARY:
This study aims to evaluate the clinical and radiological outcomes of patients undergoing anatomical single-bundle anterior cruciate ligament reconstruction with periosteal-patellar tendon-bone autograft and press-fit tibial fixation technique. The study also aims to compare these outcomes with other reconstruction techniques in the literature. The research investigates the results of a novel surgical technique, providing a minimally invasive and faster rehabilitation for patients undergoing surgery due to anterior cruciate ligament rupture. The technique does not use any screws or staples for tibial fixation, but it carries similar risks as existing techniques. The technique, similar to the well-known bone-patellar tendon-bone (BPTB) autograft technique, creates minimal bone defect at the tibial tuberosity. Over time, the defect remodels and causes minimal clinical discomfort. Despite these limitations, the authors expect patients operated with the investigated new technique to experience less postoperative swelling, less pain, faster mobilization, and earlier rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent anatomical single-bundle anterior cruciate ligament reconstruction with periosteal - patellar tendon - bone autograft and press-fit tibial fixation technique after anterior cruciate ligament rupture
* patients with at least 1 year of clinical and radiological follow-up
* patients who did not undergo a revision

Exclusion Criteria:

* Patients who underwent a secondary arthroscopy for any reason after primary surgery
* Patients with a history of septic arthritis (before and after the surgery)
* Those with a history of trauma after primary surgery to the operated knee
* Patients who have not completed at least 1 year of follow-up

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients with a diagnosis of ruptured ACL scheduled for surgery with the aforementioned technique.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2025-11-25 (Estimated); Study Completion 2025-11-25 (Estimated)

PRIMARY OUTCOMES:
The Knee injury and Osteoarthritis Outcome Score (KOOS) | Postoperative 1.st year
  minimum value:0, maximum value 100, higher values mean better outcome
The International Knee Documentation Committee Score (IKDC) | Postoperative 1.st year
  minimum value:0, maximum value 100, higher values mean better outcome
Tegner-Lysholm Scale | Postoperative 1.st year
  minimum value:0, maximum value 100, higher values mean better outcome
Graft survival | Postoperative 1.st year
  Overall graft survival

SECONDARY OUTCOMES:
Tunnel widening | Postoperative 1.st year
  Tibial and femoral tunnel widening will be measured on direct calibrated Xrays as a distance (in millimeters) and on CT scans taken at the sixth postoperative month. The distance will be measured on the widest point between the sclerotic lines on the Xrays and perpendicular to their longitudinal trajectories.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Akoto R, Muller-Hubenthal J, Balke M, Albers M, Bouillon B, Helm P, Banerjee M, Hoher J. Press-fit fixation using autologous bone in the tibial canal causes less enlargement of bone tunnel diameter in ACL reconstruction--a CT scan analysis three months postoperatively. BMC Musculoskelet Disord. 2015 Aug 19;16:200. doi: 10.1186/s12891-015-0656-5. PMID 26285568
- [Background] Barie A, Sprinckstub T, Huber J, Jaber A. Quadriceps tendon vs. patellar tendon autograft for ACL reconstruction using a hardware-free press-fit fixation technique: comparable stability, function and return-to-sport level but less donor site morbidity in athletes after 10 years. Arch Orthop Trauma Surg. 2020 Oct;140(10):1465-1474. doi: 10.1007/s00402-020-03508-1. Epub 2020 Jun 5. PMID 32504178
- [Background] Arnold MP, Burger LD, Wirz D, Goepfert B, Hirschmann MT. The biomechanical strength of a hardware-free femoral press-fit method for ACL bone-tendon-bone graft fixation. Knee Surg Sports Traumatol Arthrosc. 2017 Apr;25(4):1234-1240. doi: 10.1007/s00167-015-3960-6. Epub 2016 Jan 7. PMID 26744280
- [Background] Haberli J, Heilgemeir M, Valet S, Aiyangar A, Overes T, Henle P, Eggli S. Novel press-fit technique of patellar bone plug in anterior cruciate ligament reconstruction is comparable to interference screw fixation. Arch Orthop Trauma Surg. 2022 Aug;142(8):1963-1970. doi: 10.1007/s00402-021-04137-y. Epub 2021 Aug 30. PMID 34462826
- [Background] Kocabey Y, Yildirim C, Erden T, Kaya A. Tibial Press-Fit Fixation Technique in Anterior Cruciate Ligament Reconstruction. Arthrosc Tech. 2023 Apr 24;12(5):e737-e743. doi: 10.1016/j.eats.2023.02.001. eCollection 2023 May. PMID 37323777